CLINICAL TRIAL: NCT01405079
Title: A Randomized, Open-label Trial of Gefitinib Versus Combination of Vinorelbine Plus Platinum as Adjuvant Treatment in Pathological Stage II-IIIA(N1-N2) Non-small Cell Lung Cancer With EGFR Mutation
Brief Title: Gefitinib Versus Vinorelbine/Platinum as Adjuvant Treatment in Stage II-IIIA(N1-N2) NSCLC With EGFR Mutation
Acronym: ADJUVANT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guangdong Association of Clinical Trials (Other)
Collaborators: Guangdong Provincial People's Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Sun Yat-sen University (Other); Jilin Provincial Tumor Hospital (Other); Liaoning Cancer Hospital & Institute (Other); First Hospital of China Medical University (Other); Chinese PLA General Hospital (Other); Peking Union Medical College Hospital (Other); Peking University People's Hospital (Other); Beijing Chest Hospital (Other); 309th Hospital of Chinese People's Liberation Army (Other); Peking University Cancer Hospital & Institute (Other); Peking University First Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other); The Affiliated Hospital of Qingdao University (Other); Jiangsu Cancer Institute & Hospital (Other); The First Affiliated Hospital of Soochow University (Other); Fudan University (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other); Zhejiang Cancer Hospital (Other); Zhejiang University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Tongji Hospital (Other); West China Hospital (Other); Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, Yi-Long Wu, Dr, Guangdong Association of Clinical Trials
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTONG 1104; CTONG 1104 (Other: Chinese Thoracic Oncology Group（CTONG）)
Record Dates: First submitted 2011-07-26; First posted 2011-07-29 (Estimated); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Lung cancer; II-IIIA(N1-N2); Adjuvant treatment; EGFR mutations; Tyrosine kinase inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gefitinib (Experimental): Gefitinib 250 mg/day oral daily
  Interventions: Drug: Gefitinib
- Vinorelbine+Cisplatin (Active Comparator): Vinorelbine 25 mg/m2 intravenous infusion on day 1 and day 8, Cisplatin 75 mg/m2 on day 1 for 4 cycles
  Interventions: Drug: Vinorelbine+Cisplatin

INTERVENTIONS:
Drug: Gefitinib — Gefitinib 250 mg/day oral daily
  Other Names: Iressa
  Arms: Gefitinib
Drug: Vinorelbine+Cisplatin — Vinorelbine 25 mg/m2 intravenous infusion on day 1 and day 8, Cisplatin 75 mg/m2 on day 1 for 4 cycles
  Arms: Vinorelbine+Cisplatin

SUMMARY:
Activating somatic mutations of the tyrosine kinase domain of epidermal growth factor receptor (EGFR) have been characterized in a subset of patients with advanced NSCLC.The EGFR mutation rate was 30% in Chinese Non-small Cell Lung Cancer(NSCLC). Patients harboring these mutations in their tumors show excellent response to EGFR tyrosine kinase inhibitors (EGFR-TKIs). This randomized phase III trial is studying gefitinib to see how well it works compared to cisplatin-based chemotherapy in treating patients who have undergone surgery for stage II-IIIA(N1-N2) NSCLC with EGFR activating mutation in Asian population.

DETAILED DESCRIPTION:
Adjuvant cisplatin-based chemotherapy is recommended for routine use in patients with stages IIA, IIB, and IIIA non-small cell lung cancer (NSCLC) after complete resection. Cisplatin and vinorelbine combination is the standard of care in adjuvant setting. The BR. 19 trial reported adjuvant gefitinib after complete resection of early stage NSCLC(stage IB 49%, II 38%, III 13%) did not confer disease free survival(DFS) or overall survival(OS) advantage in overall population. While the median gefitinib treatment time is only 4.8 months. There are only 76 patients with EGFR mutations included in this analysis. The study closed prematurely in 2005.

Activating somatic mutations of the tyrosine kinase domain of epidermal growth factor receptor (EGFR) have been characterized in a subset of patients with advanced NSCLC.The EGFR mutation rate was 30% in Chinese NSCLC. Patients harboring these mutations in their tumors show excellent response to EGFR tyrosine kinase inhibitors (EGFR-TKIs). This randomized phase III trial is studying gefitinib to see how well it works compared to cisplatin-based chemotherapy in treating patients who have undergone surgery for stage II-IIIA(N1-N2) NSCLC with EGFR activating mutation in Asian population.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided.
* Males or females aged ≥18 years, < 75 years.
* Able to comply with the required protocol and follow-up procedures, and able to receive oral medications.
* Target population is completely resected pathological stage II-IIIA(N1-N2) NSCLC with EGFR exon 19 deletions and exon 21 L858R activating mutation.
* Patient who can start the investigational therapy within 3-6 weeks after the complete resection
* ECOG performance status 0-1.
* Life expectancy ≥12 weeks.
* Adequate hematological function: Absolute neutrophil count (ANC) ≥2.0 x 109/L, and Platelet count ≥100 x 109/L, and Hemoglobin ≥9 g/dL (may be transfused to maintain or exceed this level).
* Adequate liver function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN), Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 x ULN in subjects without liver metastases; ≤ 5 x ULN in subjects with liver metastases.
* Adequate renal function: Serum creatinine ≤ 1.25 x ULN, or ≥ 60 ml/min.
* Female subjects should not be pregnant or breast-feeding.

Exclusion Criteria:

* Known severe hypersensitivity to gefitinib or any of the excipients of this product.
* Known severe hypersensitivity to pre-medications required for treatment with cisplatin / vinorelbine doublet chemotherapy.
* Inability to comply with protocol or study procedures.
* A serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study.
* A serious cardiac condition, such as myocardial infarction within 6 months, angina, or heart disease.
* Interstitial pneumonia.
* Patients with prior exposure to agents directed at the HER axis (e.g. erlotinib, gefitinib, cetuximab, trastuzumab).
* Patients with prior chemotherapy or therapy with systemic anti-tumour therapy (e.g. monoclonal antibody therapy).
* Patients with prior radiotherapy
* History of another malignancy in the last 5 years with the exception of the following:Other malignancies cured by surgery alone and having a continuous disease-free interval of 5 years are permitted. Cured basal cell carcinoma of the skin and cured in situ carcinoma of the uterine cervix are permitted.
* Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).
* Eye inflammation or eye infection not fully treated or conditions predisposing the subject to this.
* Evidence of any other disease, neurological or metabolic dysfunction, physical examination or laboratory finding giving reasonable suspicion of a disease or condition that contraindicated the use of an investigational drug or puts the subject at high risk for treatment-related complications.
* Patient who has active serious infection (e.g. pyrexia of or 38.0℃ over)
* Patients who harbouring exon 20 T790M mutation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2011-09-19 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | Pts after surgery will receive long-term follow-up including chest CT scan, abdominal ultrasound every 3 months, brain MRI every 6 months, bone scan every 12 months for up to 3 years. The survival after 3 years will be followed up with telephone.
  To evaluate the disease free survival of gefitinib versus combination of vinorelbine plus platinum as adjuvant treatment for pathological stage II-IIIA(N1-N2) NSCLC with EGFR mutation.Disease free survival (DFS)- defined as the time from randomization to the first documented disease progression or death, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival | Pts after surgery will receive long-term follow-up including chest CT scan, abdominal ultrasound every 3 months, brain MRI every 6 months, bone scan every 12 months for up to 3 years. The survival after 3 years will be followed up with telephone.
  To evaluate the overall survival of gefitinib versus combination of vinorelbine plus platinum as adjuvant treatment for stage II-IIIA(N1-N2) NSCLC with EGFR mutation.
3 yeas DFS rate, 5 years DFS rate, 5 years OS rate | Pts after surgery will receive long-term follow-up including chest CT scan, abdominal ultrasound every 3 months, brain MRI every 6 months, bone scan every 12 months for up to 3 years. The survival after 3 years will be followed up with telephone.
  To compare the randomized treatment arms in terms of 3 yeas DFS rate, 5 years DFS rate, 5 years OS rate.
Number of Participants with Adverse Events | In the period of Gefitinib 250 mg/day oral daily for 24 months.Vinorelbine 25 mg/m2 intravenous infusion on day 1 and day 8, Cisplatin 75 mg/m2 on day 1 for 4 cycles.
  The safety and tolerability profile of gefitinib at a 250 mg daily dose relative to that of Chemotherapy.
The Total Score and TOI of FACT-L to Measure Quality of life | In the period of Gefitinib 250 mg/day oral daily for 24 months.Vinorelbine 25 mg/m2 intravenous infusion on day 1 and day 8, Cisplatin 75 mg/m2 on day 1 for 4 cycles.
  Quality of life as measured by the total score and Trial Outcome Index (TOI) of the Functional Assessment of Cancer Therapy - Lung Cancer (FACT-L) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Long WU, MD, Principal Investigator — Guangdong Provincial People's Hospital; Xue-Ning YANG, MD, Study Chair — Guangdong Provincial People's Hospital; Wen-Zhao ZHONG, MD, Study Director — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Janjigian YY, Park BJ, Zakowski MF, Ladanyi M, Pao W, D'Angelo SP, Kris MG, Shen R, Zheng J, Azzoli CG. Impact on disease-free survival of adjuvant erlotinib or gefitinib in patients with resected lung adenocarcinomas that harbor EGFR mutations. J Thorac Oncol. 2011 Mar;6(3):569-75. doi: 10.1097/JTO.0b013e318202bffe. PMID 21150674
- [Derived] Occhipinti M, Imbimbo M, Ferrara R, Simeon V, Fiscon G, Marchal C, Skoetz N, Viscardi G. Adjuvant epidermal growth factor receptor (EGFR) tyrosine kinase inhibitors (TKIs) for the treatment of people with resected stage I to III non-small-cell lung cancer and EGFR mutation. Cochrane Database Syst Rev. 2025 May 27;5(5):CD015140. doi: 10.1002/14651858.CD015140.pub2. PMID 40421698
- [Derived] Zhong WZ, Wang Q, Mao WM, Xu ST, Wu L, Wei YC, Liu YY, Chen C, Cheng Y, Yin R, Yang F, Ren SX, Li XF, Li J, Huang C, Liu ZD, Xu S, Chen KN, Xu SD, Liu LX, Yu P, Wang BH, Ma HT, Yang JJ, Yan HH, Yang XN, Liu SY, Zhou Q, Wu YL. Gefitinib Versus Vinorelbine Plus Cisplatin as Adjuvant Treatment for Stage II-IIIA (N1-N2) EGFR-Mutant NSCLC: Final Overall Survival Analysis of CTONG1104 Phase III Trial. J Clin Oncol. 2021 Mar 1;39(7):713-722. doi: 10.1200/JCO.20.01820. Epub 2020 Dec 17. PMID 33332190
- [Derived] Zhong WZ, Wang Q, Mao WM, Xu ST, Wu L, Shen Y, Liu YY, Chen C, Cheng Y, Xu L, Wang J, Fei K, Li XF, Li J, Huang C, Liu ZD, Xu S, Chen KN, Xu SD, Liu LX, Yu P, Wang BH, Ma HT, Yan HH, Yang XN, Zhou Q, Wu YL; ADJUVANT investigators. Gefitinib versus vinorelbine plus cisplatin as adjuvant treatment for stage II-IIIA (N1-N2) EGFR-mutant NSCLC (ADJUVANT/CTONG1104): a randomised, open-label, phase 3 study. Lancet Oncol. 2018 Jan;19(1):139-148. doi: 10.1016/S1470-2045(17)30729-5. Epub 2017 Nov 21. PMID 29174310